CLINICAL TRIAL: NCT02434276
Title: A Phase II, Multicenter, Randomized, Double-Blind, Active Comparator Controlled Study of the Immunogenicity and Safety of VAX2012Q, A Quadrivalent Influenza Vaccine in Healthy Adults 18-64 Years
Brief Title: Study of the Immunogenicity and Safety of a Quadrivalent Influenza Vaccine (VAX2012Q) in Adults 18-64 Years
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VaxInnate Corporation (Industry)
Collaborators: Accelovance (Industry); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAX2012Q-03
Record Dates: First submitted 2015-04-16; First posted 2015-05-05 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine Dose Group 8 mcg dose (Experimental): VAX2012Q, 8 mcg dose
  Interventions: Biological: VAX2012Q
- Vaccine Dose Group 12 mcg dose (Experimental): VAX2012Q, 12 mcg dose
  Interventions: Biological: VAX2012Q
- Control (Active Comparator): Fluzone Quadrivalent vaccine
  Interventions: Biological: Fluzone Quadrivalent

INTERVENTIONS:
Biological: VAX2012Q — Recombinant influenza hemagglutinin (HA) vaccine consisting of two influenza A subtypes and two influenza B lineages
  Other Names: Quadrivalent Recombinant Hemagglutinin Influenza Vaccine; RIV4
  Arms: Vaccine Dose Group 12 mcg dose; Vaccine Dose Group 8 mcg dose
Biological: Fluzone Quadrivalent — Fluzone Quadrivalent (Influenza Vaccine)
  Other Names: IIV4
  Arms: Control

SUMMARY:
This is a multi-center, randomized, double-blind, active comparator controlled study in which up to 450 healthy adults age 18-64 years will be administered either one of two dose levels of VAX2012Q or a licensed quadrivalent influenza vaccine. The subjects will be randomized at a 1:1:1 ratio.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, active comparator controlled study in which up to 450 healthy adults age 18-64 years will be administered either VAX2012Q or Fluzone. Four hundred fifty (450) subjects will be randomized 1:1:1 ratio of either 8 or 12 mcg VAX2012Q dose levels or to Fluzone® Quadrivalent vaccine.

Randomization will be stratified for age (18-49 and 50-64 years). Subjects will be stratified by two age groups (18-49 and 50-64) and randomized in a 1:1:1 ratio to either 8 or 12 mcg VAX2012Q dose levels or to Fluzone® Quadrivalent vaccine. 25-35% of the total study population will be recruited into the 50-64 age group.

The primary objective of the study is to evaluate the seroconversion rates at Day 21 for both dose levels of VAX2012Q.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-64 years of age.
* Females must be:

  1. Surgically sterilized
  2. Post menopausal:
* 12 months of spontaneous amenorrhea or
* 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 milli-International Units (mIU)/ml or
* 6 weeks postsurgical bilateral oophorectomy

  3. Those of childbearing potential must have a negative pre-treatment serum pregnancy test followed by a confirmatory urine pregnancy test immediately prior to vaccination and must agree to use a reliable form of contraception for at least 21 days post vaccination including contraceptives, intrauterine device, double-barrier method.
* In good health as determined by medical history, physical exam, laboratory assessments and the clinical judgment of the Principal Investigator.
* Must sign informed consent indicating understanding of the purpose of and procedures required for the study and willingness to participate.

Exclusion Criteria:

* Within 6 months preceding the administration of the study vaccine, receiving any licensed or investigational vaccine.
* Within 30 days preceding the administration of the study vaccine, receiving any investigational drug.
* Excessive chronic alcohol use within the last 5 years.
* History of drug abuse, other than recreational cannabis use, within the last 5 years that could affect the subject's participation in the study.
* Significant psychiatric illness within the last 12 months which would interfere with the study.
* A chronic illness that is not medically stable, receiving a concomitant therapy in which the medication dose has not been stable for at least 3 months prior to immunization or has any other condition that could interfere with the study.
* Clinically significant abnormal liver function tests at screening: alanine transaminase (ALT) or aspartate aminotransferase (AST) >2.5 Upper Limit of Normal (ULN).
* Total bilirubin > 1.5 ULN if ALT or AST > ULN or total bilirubin > 2 ULN with ALT and AST within normal range .
* Creatinine >1.7mg/dL, Hemoglobin < 11g/dL for females; <12.5 g/dL for males, white blood cells (WBC) <2500cell/mm3 or > 15,000cell/mm3, Platelet Count <125,000cell/mm3
* Positive serology for HBSAg, hepatitis C virus (HCV) or HIV
* Have cancer or have received treatment for cancer within three years, excluding in situ cervical carcinoma or basal /squamous cell carcinoma of the skin at other than the vaccination site.
* Any autoimmune disease.
* Presently receiving or having a recent history of receiving (≤ six months) any medication or therapeutic modality that affects the immune system or a drug known to be frequently associated with significant major organ toxicity or system corticosteroids (oral or injectable).
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any seasonal influenza vaccine component.
* Allergic to egg or egg products.
* History of Guillain-Barré Syndrome.
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the three week study period following vaccination
* Donation of blood or blood products within 4 weeks prior to vaccination or during the 4 week study period following vaccination.
* Acute disease within 72 hours prior to vaccination.
* An oral temperature >100.4°F (38°C) on the day of vaccination
* Body Mass Index >40.
* Known bleeding disorders or receiving prescribed oral or parenteral anticoagulants.
* Any other condition or circumstance which, in the opinion of the Principal Investigator, poses an unacceptable risk for participation in the study or could interfere with study evaluations.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rates to the 4 components of VAX2012Q | Through day 21
  Immune response to the vaccine will be measured in sera by the hemagglutination inhibition (HAI) assay.

SECONDARY OUTCOMES:
Safety following vaccination assessed by Adverse events (AEs) | Through day 21
  vital signs, laboratory test results and analgesic and antipyretic use to treat symptoms emerging post vaccination will be collected.
Immunogenicity of the two dose levels of VAX2012Q and of Fluzone Quadrivalent | Through day 21
  Immune responses to the vaccines will be measured in sera by HAI assay.
C-reactive protein levels | Through day 7
  Measure C-reactive protein levels.
Long term safety following vaccination assessed by Clinically significant AEs | After Day 21 through one year
  including Serious Adverse Events, Adverse Events of Special Interest and new onset chronic diseases, will be collected.

OTHER OUTCOMES:
Duration of immunity | Through day 90
  Immune responses will be measured in sera by HAI assay.
Breadth of immunity | Through day 90
  Immune responses to influenza virus strains not contained in the vaccines will be measured in sera by HAI assay.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Haworth, MD, Study Director — VaxInnate Corporation
Locations (6):
- United States (6):
  - Optimal Research, Huntsville, Alabama
  - Optimal Research, San Diego, California
  - Optimal Research, Melbourne, Florida
  - Optimal Research, Peoria, Illinois
  - Optimal Research, Mishawaka, Indiana
  - Optimal Research, Rockville, Maryland